CLINICAL TRIAL: NCT02032888
Title: A Phase 3 Evaluation of Daclatasvir Plus Sofosbuvir in Treatment-naïve and Treatment-experienced Chronic Hepatitis C (Genotype 1, 2, 3, 4, 5, or 6) Subjects Coinfected With Human Immunodeficiency Virus (HIV)
Brief Title: A Phase 3 Study to Evaluate Combination Therapy With Daclatasvir and Sofosbuvir in the Treatment of HIV and Hepatitis C Virus Coinfection.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AI444-216
Record Dates: First submitted 2014-01-09; First posted 2014-01-10 (Estimated); Results first posted 2015-10-27 (Estimated); Last update posted 2015-10-27 (Estimated); Status verified 2015-08

CONDITIONS: Hepatitis C
MeSH Terms: conditions — Hepatitis C | interventions — daclatasvir; Sofosbuvir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Daclatasvir + Sofosbuvir (Treatment-naive) 12 weeks (Experimental): Treatment-naïve participants received daclatasvir 30, 60, or 90 mg, and sofosbuvir, 400 mg, once daily for 12 weeks
  Interventions: Drug: Daclatasvir; Drug: Sofosbuvir
- Daclatasvir + Sofosbuvir (Treatment-naive) 8 weeks (Experimental): Treatment-naïve participants received daclatasvir, 30, 60, or 90 mg, and sofosbuvir, 400 mg, once daily for 8 weeks
  Interventions: Drug: Daclatasvir; Drug: Sofosbuvir
- Daclatasvir + Sofosbuvir (Treatment-experienced) 12 weeks (Experimental): Treatment-experienced participants received daclatasvir, 30, 60, or 90 mg, and sofosbuvir, 400 mg, once daily for 12 weeks
  Interventions: Drug: Daclatasvir; Drug: Sofosbuvir

INTERVENTIONS:
Drug: Daclatasvir
  Other Names: BMS-790052
Drug: Sofosbuvir

SUMMARY:
A study of the efficacy and safety of the combination of daclatasvir and sofosbuvir in the treatment of hepatitis C virus and HIV coinfection.

ELIGIBILITY:
For more information regarding BMS clinical trial participation, please visit www.BMSStudyConnect.com

Key Inclusion Criteria:

* Patients must be able to understand and agree to/comply with the prescribed dosing regimens and procedures, report for regularly scheduled study visits, and reliably communicate with study personnel about adverse events and concomitant medications
* Patients chronically infected with hepatitis C virus (HCV) genotype 1, 2, 3, 4, 5, or 6, as documented by positive HCV RNA at screening
* Patients who are HCV treatment-naive
* Patients who are HCV treatment-experienced and who have had prior anti-HCV therapies discontinued or completed at least 12 weeks prior to screening
* Patients with HCV RNA ≥10,000 IU/mL at screening
* Patients with HIV-1 infection

Key Exclusion Criteria:

* Presence of AIDs-defining opportunistic infections, as defined by the Centers of Disease Control and Prevention, within 12 weeks prior to study entry
* Patients infected with HIV-2
* Liver or any other organ transplant (including hematopoietic stem cell transplants) other than cornea and hair
* Current or known history of cancer (except in situ carcinoma of the cervix or adequately treated basal or squamous cell carcinoma of the skin) within 5 years prior to screening
* Documented or suspected hepatocellular carcinoma, as evidenced by previously obtained imaging studies or liver biopsy (or on a screening imaging study/liver biopsy if this was performed
* Evidence of decompensated liver disease, including radiologic criteria, a history or presence of ascites, bleeding varices, or hepatic encephalopathy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 238 (Actual)
Dates: Start 2014-02; Primary Completion 2014-10 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (37):
- United States (37):
  - University Of Alabama At Birmingham, Birmingham, Alabama
  - Pacific Oaks Medical Group, Beverly Hills, California
  - Va Long Beach Healthcare System, Long Beach, California
  - Peter J Ruane Md Inc, Los Angeles, California
  - Anthony M. Mills Md Inc, Los Angeles, California
  - Jeffrey Goodman Special Care Clinic, Los Angeles, California
  - Ucsd Antiviral Research Center (Avrc), San Diego, California
  - Precision Research Institute, Llc, San Diego, California
  - University Of California San Francisco, San Francisco, California
  - University Of Colorado, Aurora, Colorado
  - Whitman Walker Health, Washington D.C., District of Columbia
  - Medstar Washington Hospital Center, Washington D.C., District of Columbia
  - Capital Medical Associates, Washington D.C., District of Columbia
  - Midway Immunology And Research Center, Ft. Pierce, Florida
  - University Of Miami Schiff Center For Liver Diseases, Miami, Florida
  - Orlando Immunology Center, Orlando, Florida
  - Infect. Disease Specialists, Decatur, Georgia
  - Indiana University Health - University Hospital, Indianapolis, Indiana
  - Digestive Disease Associates, P.A., Baltimore, Maryland
  - Johns Hopkins University, Lutherville, Maryland
  - Henry Ford Health System, Detroit, Michigan
  - Washington University School Of Medicine, St Louis, Missouri
  - Southwest Care Center, Sante Fe, New Mexico
  - Binghamton Gastroenterology Associates, Binghamton, New York
  - Icahn School Of Medicine At Mount Sinai, New York, New York
  - University Of Cincinnati, Cincinnati, Ohio
  - Healthcare Research Consultants, Tulsa, Oklahoma
  - Oregon Health Science Univ, Portland, Oregon
  - Lehigh Valley Health Network, Allentown, Pennsylvania
  - University Gastroenterology, Providence, Rhode Island
  - The Miriam Hospital, Providence, Rhode Island
  - Tarrant County Inf Dis Assoc, Fort Worth, Texas
  - Cure C Consortium, Houston, Texas
  - University Of Texas Health Science Center At Houston, Houston, Texas
  - Clinical Research Centers Of America, Murray, Utah
  - Mcguire D V A M C, Richmond, Virginia
  - Harborview Medical Center, Seattle, Washington

REFERENCES:
- [Derived] Luetkemeyer AF, McDonald C, Ramgopal M, Noviello S, Bhore R, Ackerman P. 12 Weeks of Daclatasvir in Combination With Sofosbuvir for HIV-HCV Coinfection (ALLY-2 Study): Efficacy and Safety by HIV Combination Antiretroviral Regimens. Clin Infect Dis. 2016 Jun 15;62(12):1489-96. doi: 10.1093/cid/ciw163. Epub 2016 Mar 29. PMID 27025835
- [Derived] Wyles DL, Ruane PJ, Sulkowski MS, Dieterich D, Luetkemeyer A, Morgan TR, Sherman KE, Dretler R, Fishbein D, Gathe JC Jr, Henn S, Hinestrosa F, Huynh C, McDonald C, Mills A, Overton ET, Ramgopal M, Rashbaum B, Ray G, Scarsella A, Yozviak J, McPhee F, Liu Z, Hughes E, Yin PD, Noviello S, Ackerman P; ALLY-2 Investigators. Daclatasvir plus Sofosbuvir for HCV in Patients Coinfected with HIV-1. N Engl J Med. 2015 Aug 20;373(8):714-25. doi: 10.1056/NEJMoa1503153. Epub 2015 Jul 21. PMID 26196502
- See also: BMS clinical trial educational resource — http://www.bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 37 sites in the United States.
Pre-assignment Details: A total of 238 participants were enrolled, and 203 received treatment. Of the 35 participants who were enrolled but did not receive treatment, 2 withdrew consent, 31 no longer met study criteria, 1 was lost to follow-up, and 1 was eliminated for other reasons.
Groups:
- Treatment-naive: Daclatasvir + Sofosbuvir 12 Weeks: Participants without prior hepatitis C virus (HCV)treatment, received daclatasvir, 60 mg, and sofosbuvir, 400 mg, once daily, for 12 weeks of treatment and 24 weeks of follow-up.
- Treatment-naive: Daclatasvir + Sofosbuvir 8 Weeks: Participants without prior HCV treatment, received daclatasvir, 60 mg, and sofosbuvir, 400 mg, once daily for 8 weeks of treatment and 24 weeks of follow-up.
- Treatment-experienced: Daclatasvir + Sofosbuvir 12 Weeks: Participants with prior HCV treatment, received daclatasvir, 60 mg, and sofosbuvir, 400 mg, once daily for 12 weeks of treatment and 24 weeks of follow-up.
Period: Treatment Period
Arm/Group | Treatment-naive: Daclatasvir + Sofosbuvir 12 Weeks | Treatment-naive: Daclatasvir + Sofosbuvir 8 Weeks | Treatment-experienced: Daclatasvir + Sofosbuvir 12 Weeks
Started | 101 | 50 | 52
Completed | 99 | 48 | 52
Not Completed | 2 | 2 | 0
Not completed — Poor compliance/noncompliance | 1 | 1 | 0
Not completed — Other | 1 | 1 | 0
Period: Follow-up Period
Arm/Group | Treatment-naive: Daclatasvir + Sofosbuvir 12 Weeks | Treatment-naive: Daclatasvir + Sofosbuvir 8 Weeks | Treatment-experienced: Daclatasvir + Sofosbuvir 12 Weeks
Started | 100 (All patients who received study drug and not a nonstudy HCV therapy before treatment Week 4) | 49 (All patients who received study drug and not a nonstudy HCV therapy before treatment Week 4) | 52
Completed | 97 | 47 | 52
Not Completed | 3 | 2 | 0
Not completed — Lost to Follow-up | 1 | 1 | 0
Not completed — Death | 1 | 1 | 0
Not completed — Other | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All participants who received at least 1 dose of active study therapy.
Groups:
- Treatment-naive: Daclatasvir + Sofosbuvir 12 Weeks: Participants without prior hepatitis C virus (HCV) treatment, received daclatasvir, 60 mg, and sofosbuvir, 400 mg, once daily for 12 weeks of treatment and 24 weeks of follow-up.
- Total: Total of all reporting groups
Arm/Group | Treatment-naive: Daclatasvir + Sofosbuvir 12 Weeks | Treatment-naive: Daclatasvir + Sofosbuvir 8 Weeks | Treatment-experienced: Daclatasvir + Sofosbuvir 12 Weeks | Total
Number analyzed (Participants) | 101 | 50 | 52 | 203
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.1 (9.77) | 50.8 (9.19) | 55.7 (6.21) | 51.7 (9.12)
Age, Customized [Number; unit: participants]
  <65 years | 96 | 47 | 49 | 192
  >=65 years | 5 | 3 | 3 | 11
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 8 | 9 | 26
  Male | 92 | 42 | 43 | 177
Hepatitis C Virus RNA [Mean (Standard Deviation); unit: log10 IU/mL] | 6.50 (0.758) | 6.40 (0.71) | 6.52 (0.789) | 6.48 (0.753)
Hepatitis C Virus RNA distribution [Number; unit: participants]
  <800,000 IU/mL | 22 | 6 | 8 | 36
  ≥800,000 IU/mL | 79 | 44 | 44 | 167

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Genotype 1 Hepatitis C Virus (HCV)-Infected Treatment-naive Participants With Sustained Virologic Response at Follow-up Week 12 (SVR12)
Description: SVR12 was defined as HCV RNA <lower limit of quantitation, target detected or target not detected at follow-up Week 12. HCV RNA levels were measured by the Roche COBAS® TaqMan® HCV Test version 2.0 from the central laboratory. For participants who missed the follow-up Week 12 visit, SVR12 was imputed using the next and closest available HCV RNA measurement after the follow-up Week 12 window.
Time Frame: At follow-up Week 12
Population: All genotype 1 treatment-naive participants who received at least 1 dose of study therapy. Here, 'number of participants analyzed' (N) signifies the number of participants evaluable for this outcome measure.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- Treatment-naive: Daclatasvir + Sofosbuvir 12 Weeks: Participants without prior hepatitis C virus treatment, received daclatasvir, 60 mg, and sofosbuvir, 400 mg, once daily for 12 weeks of treatment and 24 weeks of follow-up.
Arm/Group | Treatment-naive: Daclatasvir + Sofosbuvir 12 Weeks
Number analyzed (Participants) | 83
Percentage of participants | 96.4 [89.8 to 99.2]

2. Secondary Outcome: Percentage of Hepatitis C Virus (HCV)/HIV-coinfected Treatment-naive Participants With Sustained Virologic Response at Follow-up Week 12 (SVR12)
Description: SVR12 was defined as HCV RNA<lower limit of quantitation, target detected, or target not detected, at follow-up Week 12. HCV RNA levels were measured by the Roche COBAS® TaqMan® HCV Test version 2.0 from the central laboratory. For participants who missed the follow-up Week 12 visit, SVR12 was imputed using the next and closest available HCV RNA measurement after the follow-up Week 12 window.
Time Frame: At follow-up Week 12
Population: All treatment-naive participants coinfected with genotype 1 HCV and HIV who received at least 1 dose of study therapy. Here, 'N' signifies the number of participants evaluable for this outcome measure.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- Treatment-naive: Daclatasvir + Sofosbuvir 8 Weeks: Participants without prior hepatitis C virus treatment, received daclatasvir, 60 mg, and sofosbuvir, 400 mg, once daily for 8 weeks of treatment and 24 weeks of follow-up.
Arm/Group | Treatment-naive: Daclatasvir + Sofosbuvir 8 Weeks
Number analyzed (Participants) | 41
Percentage of participants | 75.6 [59.7 to 87.6]

3. Secondary Outcome: Percentage of Hepatitis C Virus (HCV)/HIV-coinfected Treatment-experienced Participants With Sustained Virologic Response at Follow-up Week 12 (SVR12)
Description: SVR12 was defined as HCV RNA <lower limit of quantitation, target detected or target not detected, at follow-up Week 12. HCV RNA levels were measured by the Roche COBAS® TaqMan® HCV Test version 2.0 from the central laboratory. For participants who missed the follow-up Week 12 visit, SVR12 was imputed using the next and closest available HCV RNA measurement after the follow-up Week 12 window.
Time Frame: At follow-up Week 12
Population: All treatment-experienced participants coinfeted with HCV/HIV who received at least 1 dose of study therapy. Here, 'N' signifies the number of participants evaluable for this outcome measure.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- Treatment-experienced: Daclatasvir + Sofosbuvir 12 Weeks: Participants with prior hepatitis C virus treatment, received daclatasvir, 60 mg, and sofosbuvir, 400 mg, once daily for 12 weeks of treatment and 24 weeks of follow-up.
Arm/Group | Treatment-experienced: Daclatasvir + Sofosbuvir 12 Weeks
Number analyzed (Participants) | 44
Percentage of participants | 97.7 [88.0 to 99.9]

4. Secondary Outcome: Percentage of Participants of All Genotypes Coinfected With Hepatitis C Virus (HCV)/HIV Who Achieved Sustained Virologic Response Rate at Follow-up Week 12 (SVR12)
Description: SVR12 was defined as HCV RNA levels <lower limit of quantitation, target detected or target not detected. HCV RNA levels were measured by the Roche COBAS® TaqMan® HCV Test version 2.0 from the central laboratory. For participants who missed the follow-up Week 12 visit, SVR12 was imputed using the next and closest available HCV RNA measurement after the follow-up Week 12 window.
Time Frame: At follow-up Week 12
Population: All participants who received at least 1 dose of study drug.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- Treatment-naive: Daclatasvir + Sofosbuvir 12 Weeks: Participants without prior hepatitis C virus (HCV)treatment received daclatasvir, 60 mg, and sofosbuvir, 400 mg, once daily for 12 weeks of treatment and 24 weeks of follow-up.
- Treatment-naive: Daclatasvir + Sofosbuvir 8 Weeks: Participants without prior HCV treatment received daclatasvir, 60 mg, and sofosbuvir, 400 mg, once daily for 8 weeks of treatment and 24 weeks of follow-up.
- Treatment-experienced: Daclatasvir + Sofosbuvir 12 Weeks: Participants with prior HCV treatment received daclatasvir, 60 mg, and sofosbuvir, 400 mg, once daily for 12 weeks of treatment and 24 weeks of follow-up.
Arm/Group | Treatment-naive: Daclatasvir + Sofosbuvir 12 Weeks | Treatment-naive: Daclatasvir + Sofosbuvir 8 Weeks | Treatment-experienced: Daclatasvir + Sofosbuvir 12 Weeks
Number analyzed (Participants) | 101 | 50 | 52
Percentage of participants | 97.0 [91.6 to 99.4] | 76.0 [61.8 to 86.9] | 98.1 [89.7 to 100]

5. Secondary Outcome: Percentage of Participants Who Achieve Hepatitis C Virus RNA Levels to be <Lower Limit of Quantitation, Target Detected (TD)or Target Not Detected (TND) at Weeks: 1, 2, 4, 6, 8, and 12; at End of Treatment; and at Follow-up Weeks 4 and 24
Description: Participants with hepatitis C virus CV) levels to be <lower limit of quantitation, TD or TND at each visit. HCV RNA levels were measured by the Roche COBAS® TaqMan® HCV Test version 2.0 from the central laboratory.
Time Frame: Week 1, 2, 4, 6, 8, 12, End of treatment, and follow-up Week 4 and 24
Population: All participants who received at least 1 dose of study drug
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- Treatment-naive: Daclatasvir + Sofosbuvir 12 Weeks: Participants without prior hepatitis C virus treatment, received daclatasvir 60-mg and sofosbuvir 400-mg OD orally, for 12 weeks of treatment and 24 weeks of follow-up.
- Treatment-naive: Daclatasvir + Sofosbuvir 8 Weeks: Participants without prior hepatitis C virus treatment, received daclatasvir 60-mg and sofosbuvir 400-mg OD orally, for 8 weeks of treatment and 24 weeks of follow-up.
- Treatment-experienced: Daclatasvir + Sofosbuvir 12 Weeks: Participants with prior hepatitis C virus treatment, received daclatasvir 60-mg and sofosbuvir 400-mg OD orally, for 12 weeks of treatment and 24 weeks of follow-up.
Arm/Group | Treatment-naive: Daclatasvir + Sofosbuvir 12 Weeks | Treatment-naive: Daclatasvir + Sofosbuvir 8 Weeks | Treatment-experienced: Daclatasvir + Sofosbuvir 12 Weeks
Number analyzed (Participants) | 101 | 50 | 52
Percentage of participants
  Week 1 | 34.7 [25.5 to 44.8] | 44.0 [30.0 to 58.7] | 34.6 [22.0 to 49.1]
  Week 2 | 77.2 [67.8 to 85.0] | 78.0 [64.0 to 88.5] | 71.2 [56.9 to 82.9]
  Week 4 | 93.1 [86.2 to 97.2] | 98.0 [89.4 to 99.9] | 92.3 [81.5 to 97.9]
  Week 6 | 99.0 [94.6 to 100.0] | 98.0 [89.4 to 99.9] | 98.1 [89.7 to 100.0]
  Week 8 | 98.0 [93.0 to 99.8] | 96.0 [86.3 to 99.5] | 100.0 [93.2 to 100.0]
  Week 12 | 96.0 [90.2 to 98.9] | NA [NA to NA] — Protocol-defined treatment duration for this arm is 8 weeks. | 98.1 [89.7 to 100.0]
  End of treatment | 99.0 [94.6 to 100.0] | 100.0 [92.9 to 100.0] | 100.0 [93.2 to 100.0]
  Follow-up Week 4 | 98.0 [93.0 to 99.8] | 82.0 [68.6 to 91.4] | 96.2 [86.8 to 99.5]
  Follow-up Week 24 | 92.1 [85.0 to 96.5] | 72.0 [57.5 to 83.8] | 92.3 [81.5 to 97.9]

6. Secondary Outcome: Percentage of Participants Coinfected With Hepatitis C Virus/HIV Who Achieved HCV RNA Levels<Lower Limit of Quantitation (LLOQ), Target Not Detected (TND)
Description: Participants with HCV RNA levels <LLOQ, TND. HCV RNA levels were measured by the Roche COBAS® TaqMan® HCV Test version 2.0 from the central laboratory.
Time Frame: At Weeks 1, 2, 4, 6, 8, and 12 and at End of Treatment
Population: All participants who received at least 1 dose of study drug
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Treatment-naive: Daclatasvir + Sofosbuvir 12 Weeks | Treatment-naive: Daclatasvir + Sofosbuvir 8 Weeks | Treatment-experienced: Daclatasvir + Sofosbuvir 12 Weeks
Number analyzed (Participants) | 101 | 50 | 52
Percentage of participants
  Week 1 | 9.9 [4.9 to 17.5] | 6.0 [1.3 to 16.5] | 5.8 [1.2 to 15.9]
  Week 2 | 33.7 [24.6 to 43.8] | 34.0 [21.2 to 48.8] | 23.1 [12.5 to 36.8]
  Week 4 | 70.3 [60.4 to 79.0] | 78.0 [64.0 to 88.5] | 63.5 [49.0 to 76.4]
  Week 6 | 89.1 [81.3 to 94.4] | 90.0 [78.2 to 96.7] | 94.2 [84.1 to 98.8]
  Week 8 | 98.0 [93.0 to 99.8] | 96.0 [86.3 to 99.5] | 100.0 [93.2 to 100.0]
  Week 12 | 96.0 [90.2 to 99.8] | NA [NA to NA] — Protocol-defined treatment duration for this arm is 8 weeks | 98.1 [89.7 to 100.0]
  End of treatment | 99.0 [94.6 to 100.0] | 100.0 [92.9 to 100.0] | 100.0 [93.2 to 100.0]

7. Secondary Outcome: Percentage of Participants With CC or Non-CC Genotype at the IL28B rs12979860 Single Nucleotide Polymorphisms Who Achieved Sustained Virologic Response at Follow-up Week 12 (SVR12)
Description: SVR is defined as hepatitis C virus RNA <lower limit of quantitation, target detected or target not detected at follow-up Week 12. Percentage calculated as number of responders/number of patients receiving treatment.
Time Frame: At Follow-up Week 12
Population: All participants who received at least 1 dose of study drug. n=participants with CC or non-CC Genotype.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- Treatment-experienced: Daclatasvir + Sofosbuvir 12 Weeks: Participants with prior HCV treatment, received daclatasvir, 60 mg, and sofosbuvi,r 400 mg, once daily for 12 weeks of treatment and 24 weeks of follow-up.
Arm/Group | Treatment-naive: Daclatasvir + Sofosbuvir 12 Weeks | Treatment-naive: Daclatasvir + Sofosbuvir 8 Weeks | Treatment-experienced: Daclatasvir + Sofosbuvir 12 Weeks
Number analyzed (Participants) | 101 | 50 | 52
Percentage of participants
  CC Genotype (n=28,13,13) | 100.0 [87.7 to 100.0] | 69.2 [38.6 to 90.9] | 100.0 [75.3 to 100.0]
  Non-CC Genotype (n=73,37, 39) | 95.9 [88.5 to 99.1] | 78.4 [61.8 to 90.2] | 97.4 [86.5 to 99.9]

8. Secondary Outcome: Number of Participants With Adverse Events (AEs), Serious Adverse Events (SAEs), AEs Leading to Interruption or Discontinuation, Treatment-related AEs/SAEs and Grade 3 to 4 AEs/SAEs and Who Died During Treatment Period
Description: AE was defined as any new unfavorable symptom, sign, or disease or worsening of a preexisting condition that may or may not have a causal relationship with treatment. SAE was defined as a medical event that at any dose resulted in death, persistent or significant disability/incapacity, or drug dependency/abuse; was life-threatening, an important medical event, or a congenital anomaly/birth defect; or required or prolonged hospitalization. AEs were categorized as Grade (Gr) 1=Mild, Gr 2=Moderate, Gr 3=Severe, Gr 4=Life-threatening or disabling, Gr 5=Death.
Time Frame: AEs: Day 1 to 7 days after last dose of study treatment (8 weeks or 12 weeks). SAEs: Day 1 to 30 days after last dose of study treatment (8 weeks or 12 weeks)
Population: All participants who received at least 1 dose of study drug.
Measure: Number; unit: Participants
Arm/Group | Treatment-naive: Daclatasvir + Sofosbuvir 12 Weeks | Treatment-naive: Daclatasvir + Sofosbuvir 8 Weeks | Treatment-experienced: Daclatasvir + Sofosbuvir 12 Weeks
Number analyzed (Participants) | 101 | 50 | 52
Participants
  AEs | 75 | 29 | 37
  SAEs | 1 | 0 | 3
  AEs requiring dose interruption or discontinuation | 0 | 0 | 0
  Treatment-related AEs | 39 | 13 | 17
  Treatment-related Grade 3 to 4 AEs | 0 | 1 | 0
  Grade 3 to 4 AEs | 3 | 2 | 4
  Death | 0 | 0 | 0

9. Secondary Outcome: Number of Participants With Adverse Events (AEs), Serious Adverse Events (SAEs), Treatment-related AEs/SAEs, Grade 3 to 4 AEs/SAEs, and Who Died During Follow-up Period
Description: as for outcome 8
Time Frame: AEs: Day 1 of follow-up period (Week 9 or Week 13) to 7 days after end of 24 weeks follow-up period. SAEs: Day 1 of follow-up period (Week 9 or Week 13) to 30 days after end of 24 weeks follow-up period.
Population: All participants who received at least 1 dose of study drug
Measure: Number; unit: Participants
Arm/Group | Treatment-naive: Daclatasvir + Sofosbuvir 12 Weeks | Treatment-naive: Daclatasvir + Sofosbuvir 8 Weeks | Treatment-experienced: Daclatasvir + Sofosbuvir 12 Weeks
Number analyzed (Participants) | 101 | 49 | 52
Participants
  AEs | 11 | 5 | 5
  SAEs | 3 | 1 | 0
  AEs Grade 3 to 4 | 3 | 1 | 0
  SAEs Grade 3 to 4 | 2 | 1 | 0
  Death | 1 | 1 | 0

10. Secondary Outcome: Number of Participants With Treatment-emergent Grade 3-4 Abnormalities on Laboratory Test Results
Description: Grade 3-4 abnormalities on laboratory test results were defined as: International normalized ratio as 2.1-3.0*upper limit of normal (ULN) for grade 3 and >3.0*ULN for grade 4. Leukocytes as 1.0*10^9-1.5*10^9/L for grade 3 and <1.0*10^9/L for grade 4. Aspartate aminotransferase as 5.1-10.0*ULN for grade 3 and >10.0*ULN for grade 4. Bilirubin (total) as 2.6-5.0*ULN for grade 3 and >5.0*ULN for grade 4. Lipase (total) as 3.1-5.0*ULN for grade 3 and >5.0*ULN for grade 4. Alanine aminotransferase as 5.1-10.0*ULN for grade 3 and >10.0*ULN for grade 4.
Time Frame: From screening up to week 24 of post treatment follow--up
Population: All participants who received at least 1 dose of study drug
Measure: Number; unit: Participants
Arm/Group | Treatment-naive: Daclatasvir + Sofosbuvir 12 Weeks | Treatment-naive: Daclatasvir + Sofosbuvir 8 Weeks | Treatment-experienced: Daclatasvir + Sofosbuvir 12 Weeks
Number analyzed (Participants) | 101 | 50 | 52
Participants
  International normalized ratio | 1 | 0 | 1
  Leukocytes | 0 | 0 | 1
  Aspartate aminotransferase | 0 | 1 | 1
  Bilirubin (total) | 5 | 1 | 2
  Lipase (total) | 5 | 1 | 1
  Alanine aminotransferase | 0 | 1 | 1

ADVERSE EVENTS:
Time Frame: AEs: From first dose of study drug to 7 days after last dose. SAEs: From baseline to 30 days after last dose of study drug
Description: On-treatment period
Arm/Group | Treatment-naive: Daclatasvir + Sofosbuvir 12 Weeks | Treatment-naive: Daclatasvir + Sofosbuvir 8 Weeks | Treatment-experienced: Daclatasvir + Sofosbuvir 12 Weeks
Serious Adverse Events (participants affected / at risk) | 1/101 | 0/50 | 3/52
Other Adverse Events (participants affected / at risk) | 51/101 | 14/50 | 25/52
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment-naive: Daclatasvir + Sofosbuvir 12 Weeks (N=101) | Treatment-naive: Daclatasvir + Sofosbuvir 8 Weeks (N=50) | Treatment-experienced: Daclatasvir + Sofosbuvir 12 Weeks (N=52)
Drug abuse (Psychiatric disorders) | 0 | 0 | 1
Hypertensive crisis (Vascular disorders) | 0 | 0 | 1
Chest pain (General disorders) | 0 | 0 | 1
Syncope (Nervous system disorders) | 0 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Presyncope (Nervous system disorders) | 0 | 0 | 1
Priapism (Reproductive system and breast disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment-naive: Daclatasvir + Sofosbuvir 12 Weeks (N=101) | Treatment-naive: Daclatasvir + Sofosbuvir 8 Weeks (N=50) | Treatment-experienced: Daclatasvir + Sofosbuvir 12 Weeks (N=52)
Dizziness (Nervous system disorders) | 1 | 2 | 3
Vomiting (Gastrointestinal disorders) | 6 | 1 | 3
Nausea (Gastrointestinal disorders) | 14 | 4 | 8
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 3 | 1
Diarrhoea (Gastrointestinal disorders) | 11 | 1 | 3
Headache (Nervous system disorders) | 12 | 3 | 8
Insomnia (Psychiatric disorders) | 5 | 0 | 3
Constipation (Gastrointestinal disorders) | 3 | 0 | 3
Fatigue (General disorders) | 19 | 5 | 10
Rash (Skin and subcutaneous tissue disorders) | 6 | 0 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.